CLINICAL TRIAL: NCT00392457
Title: Feedback Control of FSH Secretion in the Human Male
Brief Title: Investigating the Regulation of Reproductive Hormones in Adult Men
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: William F. Crowley Jr., MD, MGH
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: R01 HD15788 - 234; R01HD015788 (NIH)
Record Dates: First submitted 2006-10-25; First posted 2006-10-26 (Estimated); Last update posted 2015-02-16 (Estimated); Status verified 2010-04

CONDITIONS: Kallmann Syndrome; Hypogonadism; Gonadal Disorder
Keywords: Idiopathic Hypogonadotropic Hypogonadism; Kallmann Syndrome; Agonadal
MeSH Terms: conditions — Kallmann Syndrome; Hypogonadism; Gonadal Disorders; Idiopathic Hypogonadotropic Hypogonadism | interventions — Ketoconazole; Gonadotropin-Releasing Hormone

INTERVENTIONS:
Drug: ketoconazole — loading dose of 1g followed by a maintenance dose of 400 mg PO QID for 7 days
Drug: gonadotropin releasing hormone (GnRH) — Pulsatile GnRH (25 ng/kg per bolus every two hours via microinfusion pump titrated to reach normal serum testosterone levels)

SUMMARY:
The purpose of the research study is to learn more about the regulation of reproductive hormones in adult men. We would like to understand what role testosterone and estradiol play in controlling the release of LH (lutenizing hormone) and FSH (follicle stimulating hormone). Testosterone and estradiol come from the testes, and LH and FSH are released from a gland in the head called the pituitary.

Men involved in the study will have detailed evaluations that involve overnight stays in the hospital and frequent blood sampling. The men in the study will also be receiving medications that affect the levels of various hormones in the body. This will allow the researchers to learn how various hormones influence each other. Men that participate in the study will receive medical evaluations and monetary compensation. Information gathered from this study will help in the development of new treatments for infertility and potentially new hormonal forms of contraception.

DETAILED DESCRIPTION:
In the United States 10-15% couples seek evaluation for infertility, of whom a male factor is identified in approximately 50% of cases. To date, however, most infertility research has focused on the female partner and in the majority of instances the etiology of male infertility remains poorly understood with inconsistent elevation in FSH levels. Given that spermatogenesis is highly dependent on FSH secretion, this project will focus on delineating the feedback control of FSH in the human male. Such studies, although difficult to perform in the human, are critical to understanding not only the pathophysiology of male infertility, but also to determining the feasibility of hormonal approaches to male contraception. In this protocol, studies of normal, GnRH-deficient and agonadal men employing reversible sex steroid ablation, physiologic sex steroid replacement and manipulation of the GnRH input to the pituitary will permit the non-steroidal, sex steroid, and GnRH-dependent components of FSH regulation to be selectively elucidated.

ELIGIBILITY:
Inclusion Criteria:

* Men aged 18 to 50 years
* In good health
* On no medications

Exclusion Criteria:

Subjects will not be enrolled in this study if there is a history of:

* Liver disease or if screening blood tests demonstrate abnormal liver function tests
* Excessive alcohol consumption
* Illicit drug use
* Severe drug allergy
* Use of any concomitant medications
* Peptic ulcer disease or gastritis

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 175 (Estimated)
Dates: Start 1995-07; Primary Completion 2007-02 (Actual); Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
serum hormone levels | Baseline, Day 3, and Day 6

CONTACTS AND LOCATIONS:
Overall Officials: William F Crowley, Jr., MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Background] Howards SS. Treatment of male infertility. N Engl J Med. 1995 Feb 2;332(5):312-7. doi: 10.1056/NEJM199502023320507. No abstract available. PMID 7816068
- [Background] Ying SY. Inhibins, activins, and follistatins: gonadal proteins modulating the secretion of follicle-stimulating hormone. Endocr Rev. 1988 May;9(2):267-93. doi: 10.1210/edrv-9-2-267. PMID 3136011
- [Background] Khoury RH, Wang QF, Crowley WF Jr, Hall JE, Schneyer AL, Toth T, Midgley AR Jr, Sluss PM. Serum follistatin levels in women: evidence against an endocrine function of ovarian follistatin. J Clin Endocrinol Metab. 1995 Apr;80(4):1361-8. doi: 10.1210/jcem.80.4.7714112.
- [Background] Hayes FJ, Hall JE, Boepple PA, Crowley WF Jr. Clinical review 96: Differential control of gonadotropin secretion in the human: endocrine role of inhibin. J Clin Endocrinol Metab. 1998 Jun;83(6):1835-41. doi: 10.1210/jcem.83.6.4884. PMID 9626105
- [Background] Santen RJ. Is aromatization of testosterone to estradiol required for inhibition of luteinizing hormone secretion in men? J Clin Invest. 1975 Dec;56(6):1555-63. doi: 10.1172/JCI108237. PMID 1104659
- [Background] Winters SJ, Janick JJ, Loriaux DL, Sherins RJ. Studies on the role of sex steroids in the feedback control of gonadotropin concentrations in men. II. Use of the estrogen antagonist, clomiphene citrate. J Clin Endocrinol Metab. 1979 Feb;48(2):222-7. doi: 10.1210/jcem-48-2-222. No abstract available. PMID 372203
- [Background] Matsumoto AM, Bremner WJ. Modulation of pulsatile gonadotropin secretion by testosterone in man. J Clin Endocrinol Metab. 1984 Apr;58(4):609-14. doi: 10.1210/jcem-58-4-609. PMID 6421864
- [Background] Finkelstein JS, Whitcomb RW, O'Dea LS, Longcope C, Schoenfeld DA, Crowley WF Jr. Sex steroid control of gonadotropin secretion in the human male. I. Effects of testosterone administration in normal and gonadotropin-releasing hormone-deficient men. J Clin Endocrinol Metab. 1991 Sep;73(3):609-20. doi: 10.1210/jcem-73-3-609. PMID 1908484
- [Background] Finkelstein JS, O'Dea LS, Whitcomb RW, Crowley WF Jr. Sex steroid control of gonadotropin secretion in the human male. II. Effects of estradiol administration in normal and gonadotropin-releasing hormone-deficient men. J Clin Endocrinol Metab. 1991 Sep;73(3):621-8. doi: 10.1210/jcem-73-3-621. PMID 1908485
- [Background] Bagatell CJ, Dahl KD, Bremner WJ. The direct pituitary effect of testosterone to inhibit gonadotropin secretion in men is partially mediated by aromatization to estradiol. J Androl. 1994 Jan-Feb;15(1):15-21. PMID 8188534
- [Background] Groome NP, Illingworth PJ, O'Brien M, Pai R, Rodger FE, Mather JP, McNeilly AS. Measurement of dimeric inhibin B throughout the human menstrual cycle. J Clin Endocrinol Metab. 1996 Apr;81(4):1401-5. doi: 10.1210/jcem.81.4.8636341.
- [Background] Majumdar SS, Mikuma N, Ishwad PC, Winters SJ, Attardi BJ, Perera AD, Plant TM. Replacement with recombinant human inhibin immediately after orchidectomy in the hypophysiotropically clamped male rhesus monkey (Macaca mulatta) maintains follicle-stimulating hormone (FSH) secretion and FSH beta messenger ribonucleic acid levels at precastration values. Endocrinology. 1995 May;136(5):1969-77. doi: 10.1210/endo.136.5.7720645.
- [Background] Culler MD, Negro-Vilar A. Passive immunoneutralization of endogenous inhibin: sex-related differences in the role of inhibin during development. Mol Cell Endocrinol. 1988 Aug;58(2-3):263-73. doi: 10.1016/0303-7207(88)90163-3. PMID 3145231
- [Background] Veldhuis JD, Johnson ML. Cluster analysis: a simple, versatile, and robust algorithm for endocrine pulse detection. Am J Physiol. 1986 Apr;250(4 Pt 1):E486-93. doi: 10.1152/ajpendo.1986.250.4.E486. PMID 3008572
- [Background] Heel RC, Brogden RN, Carmine A, Morley PA, Speight TM, Avery GS. Ketoconazole: a review of its therapeutic efficacy in superficial and systemic fungal infections. Drugs. 1982 Jan-Feb;23(1-2):1-36. doi: 10.2165/00003495-198223010-00001. No abstract available. PMID 6276122
- [Background] Pont A, Graybill JR, Craven PC, Galgiani JN, Dismukes WE, Reitz RE, Stevens DA. High-dose ketoconazole therapy and adrenal and testicular function in humans. Arch Intern Med. 1984 Nov;144(11):2150-3. PMID 6093722
- [Background] Sonino N. The use of ketoconazole as an inhibitor of steroid production. N Engl J Med. 1987 Sep 24;317(13):812-8. doi: 10.1056/NEJM198709243171307. No abstract available. PMID 3306384
- [Background] Van Tyle JH. Ketoconazole. Mechanism of action, spectrum of activity, pharmacokinetics, drug interactions, adverse reactions and therapeutic use. Pharmacotherapy. 1984 Nov-Dec;4(6):343-73. doi: 10.1002/j.1875-9114.1984.tb03398.x. PMID 6151171
- [Background] Lewis JH, Zimmerman HJ, Benson GD, Ishak KG. Hepatic injury associated with ketoconazole therapy. Analysis of 33 cases. Gastroenterology. 1984 Mar;86(3):503-13. PMID 6319220
- [Background] Duarte PA, Chow CC, Simmons F, Ruskin J. Fatal hepatitis associated with ketoconazole therapy. Arch Intern Med. 1984 May;144(5):1069-70. PMID 6324708
- [Background] van Dijke CP, Veerman FR, Haverkamp HC. Anaphylactic reactions to ketoconazole. Br Med J (Clin Res Ed). 1983 Dec 3;287(6406):1673. doi: 10.1136/bmj.287.6406.1673. No abstract available. PMID 6315129
- [Background] Janssen PA, Symoens JE. Hepatic reactions during ketoconazole treatment. Am J Med. 1983 Jan 24;74(1B):80-5. doi: 10.1016/0002-9343(83)90519-3. PMID 6129799
- [Result] Pitteloud N, Dwyer AA, DeCruz S, Lee H, Boepple PA, Crowley WF Jr, Hayes FJ. Inhibition of luteinizing hormone secretion by testosterone in men requires aromatization for its pituitary but not its hypothalamic effects: evidence from the tandem study of normal and gonadotropin-releasing hormone-deficient men. J Clin Endocrinol Metab. 2008 Mar;93(3):784-91. doi: 10.1210/jc.2007-2156. Epub 2007 Dec 11. PMID 18073301
- [Result] Boepple PA, Hayes FJ, Dwyer AA, Raivio T, Lee H, Crowley WF Jr, Pitteloud N. Relative roles of inhibin B and sex steroids in the negative feedback regulation of follicle-stimulating hormone in men across the full spectrum of seminiferous epithelium function. J Clin Endocrinol Metab. 2008 May;93(5):1809-14. doi: 10.1210/jc.2007-2450. Epub 2008 Feb 12. PMID 18270253
- [Result] Pitteloud N, Dwyer AA, DeCruz S, Lee H, Boepple PA, Crowley WF Jr, Hayes FJ. The relative role of gonadal sex steroids and gonadotropin-releasing hormone pulse frequency in the regulation of follicle-stimulating hormone secretion in men. J Clin Endocrinol Metab. 2008 Jul;93(7):2686-92. doi: 10.1210/jc.2007-2548. Epub 2008 Apr 29. PMID 18445673
- See also: Clinical research studies of the Reproductive Endocrine Unit at the Massachusetts General Hospital. Click here for more information about this study: Feedback Control of FSH Secretion in the Human Male — http://www.massgeneral.org/reproendo/pages/reu_study_subject.htm